CLINICAL TRIAL: NCT02860390
Title: Denver Health Asthma Management Program
Acronym: DHAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-0308 (Anderson)
Record Dates: First submitted 2016-08-03; First posted 2016-08-09 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Adolescent - Control (No Intervention): Usual care arm of subjects aged 13-19 years old
- Adolescent - SMS (Experimental): Subjects aged 13-19 years and receiving Denver Health Asthma Management Program (text messaging intervention)
  Interventions: Other: Denver Health Asthma Management Program
- Adolescent - SMS plus support person (Experimental): Subjects aged 13-19 years, Denver Health Asthma Management Program (text messaging intervention) sent to subjects and subjects' chosen Person of Support.
  Interventions: Other: Denver Health Asthma Management Program; Other: Person of Support
- Adult - Control (No Intervention): Usual care arm of subjects aged 20-40 years old.
- Adult - SMS (Experimental): Subjects aged 20-40 years and receiving Denver Health Asthma Management Program (text messaging intervention).
  Interventions: Other: Denver Health Asthma Management Program

INTERVENTIONS:
Other: Denver Health Asthma Management Program — text message (SMS) support including educational, motivational, and resource content.
  Arms: Adolescent - SMS; Adolescent - SMS plus support person; Adult - SMS
Other: Person of Support — Subjects in the adolescent cohort will designate a support person (e.g. parent) to receive messages from the Denver Health Asthma Management Program
  Arms: Adolescent - SMS plus support person

SUMMARY:
This is a Comparison Effectiveness Research (CER) study in a population of 13 to 40 year-old individuals with persistent asthma comparing differing levels of texting interventions with each other and with a usual care group. The two texting interventions include 1) texting only the individual with asthma and 2) texting the individual with asthma and an important person in that individual's life such as a parent or spouse. These two texting groups will be compared to a group receiving usual asthma care at Denver Health.

DETAILED DESCRIPTION:
This is Phase 2 of a two-phase pilot project to build and study a texting program for patients at Denver Health who have persistent asthma. The overall goal of the program is to provide educational support for asthma care between clinic visits and to survey for evidence of poorly controlled asthma, which would prompt clinic recall. Phase 1 used a focus group/interview methodology to inform Phase 2 and allow Phase 2 to be more patient-centered. Based on results of focus groups/interviews, the investigators will conduct a three-arm trial among 13- to 19-year-olds and a two-arm trial among 20- to 40-year-olds. For the 13- to 19-year-old group, a 'usual care' group will be compared to two intervention groups: 1) a subject group receiving text messages about asthma care and 2) a group of subjects and their 'significant other', such as a parent, who will also receive the text messages. Overall, Phase 1 findings suggested the 20- to 40-year-old group was more reluctant to involve a significant other and therefore for this group a 'usual care' arm will be compared to an arm where only the patient receives the text messages, but not a significant other. Other features built into Phase 2 upon recommendation from the focus group/interview phase include a midpoint survey and tailoring the amount of texting a patient receives based on the level of asthma control elicited by administration of the validated tool, the Asthma Control Test (ACT).

ELIGIBILITY:
Inclusion Criteria:

* Subject and significant other as applicable must have phone or other device capable of receiving text messages
* Ages 13 to 19 with persistent asthma per Denver Health electronic health record and/or HEDIS (modified) criteria for asthma
* Ages 20 to 40 with HEDIS (modified) criteria for persistent asthma
* Hospital-based utilization for asthma (i.e. persistent asthma)
* Denver Health Primary Care Provider visits within last 3 years
* Ability to read English or Spanish.

Exclusion Criteria:

* complex and special health care needs pediatric patients
* pregnant/expectant mothers
* incarcerated individuals
* Non-English and non-Spanish speakers
* Chronic Obstructive Pulmonary Disease/COPD or other non-asthma pulmonary diagnoses (e.g. pulmonary function testing inconsistent with asthma and/or negative methacholine challenge testing/lack of reversibility with β-agonist, diagnostic errors despite inclusion in the Asthma Registry)
* Patients who by input of the primary care provider are less likely to participate in an interactive asthma text messaging trial (e.g. intellectual delay, mental health issues)

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 154 (Actual)
Dates: Start 2016-05; Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Mean Asthma Control Test Score | Six months

SECONDARY OUTCOMES:
Asthma-related utilization - Emergent Care | Six months
  Emergent care
Asthma-related utilization - Urgent Care | Six months
  Urgent Care
Asthma-related utilization - Hospitalization | Six months
  Hospitalizations
Quality of Life | Six months
  as measured by the Juniper Asthma Quality of Life Questionnaire(s) and PHQ-4
Medication Adherence | Six months
  as measured by the Asthma Medication Ratio
Pre/Post Comparison of Asthma Control Test score | Six months

IPD SHARING:
Plan to Share IPD: No